CLINICAL TRIAL: NCT05185960
Title: Comparison of the Postprandial Glycemic and Insulinemic Response of ALLSWEET When Taken Alone or When Added to Sucrose: A Randomized, Double Blind, Controlled Clinical Trial in Healthy Individuals
Brief Title: Comparison of the Postprandial Glycemic and Insulinemic Response of ALLSWEET When Taken Alone or When Added to Sucrose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Advanced Ingredients (Industry)
Collaborators: INQUIS Clinical Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: INQ-2117
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Blood Sugar
MeSH Terms: interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ALLSWEET® (Experimental): ALLSWEET® will be mixed with 250ml of water and an additional 125ml of water. Fingerprick blood samples will be taken for 2 hours following consumption of beverage in order to assess the glycemic response.
  Interventions: Other: ALLSWEET®
- ALLSWEET® consumed with sucrose (Experimental): ALLSWEET® and sucrose will be mixed with 250ml of water and an additional 125ml of water. Fingerprick blood samples will be taken for 2 hours following consumption of beverage in order to assess the glycemic response.
  Interventions: Other: ALLSWEET® and sucrose
- Sucrose (Active Comparator): Sucrose will be mixed with 250ml of water and an additional 125ml of water. Fingerprick blood samples will be taken for 2 hours following consumption of beverage in order to assess the glycemic response.
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: ALLSWEET® — ALLSWEET®, is a non-GMO certified allulose developed by the study sponsor. It will be diluted in water.
  Arms: ALLSWEET®
Other: ALLSWEET® and sucrose — ALLSWEET®, is a non-GMO certified allulose developed by the study sponsor. It will be added to sucrose (table sugar) and diluted in water.
  Arms: ALLSWEET® consumed with sucrose
Other: Sucrose — Table sugar. It will be consumed by diluting it in water.
  Arms: Sucrose

SUMMARY:
This study will explore the postprandial glycemic response of ALLSWEET®, a non-GMO certified allulose, when consumed alone or with sucrose, compared to the consuming sucrose alone. On 3 separate days, subjects will consume in random order ALLSWEET® alone, ALLSWEET® added to sucrose, or sucrose alone. Blood samples for glucose and insulin analysis with be taken for 2 hours following consumption of the beverages.

DETAILED DESCRIPTION:
Each subject will receive 3 test meals in a double blinded, randomized, crossover fashion.

1. Test arm 1: 30g sucrose
2. Test arm 2: 30g sucrose + 15g of ALLSWEET®
3. Test arm 3: 15g ALLSWEET® All sweeteners will be mixed with 250ml of water.

Eligible subjects will be studied on 3 separate days over a period of 4 weeks or less, with at least 1 day in between test days. A fasting fingerprick blood sample will be collected for glucose and insulin analysis after which the test meal will be administered. Additional fingerprick blood samples will be drawn over the next 2 hours (15', 30', 45', 60', 90' and 120' after the first sip of the test drink).

Power calculation: A sample size of 15 subjects, is sufficient to detect a 25% difference in incremental area under the curve between meals with 80% statistical power.

Statistical Analysis: Incremental area under the curve values, blood glucose and insulin concentrations and increments at each time will be subjected to repeated-measures analysis of variance. After demonstration of significant heterogeneity, the significance of the differences between individual means will be assessed using Tukey's test to adjust for multiple comparisons, with the criterion for significance being two-tailed p<0.05. Means which differ by more than the least significant difference differ significantly.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, 20-70 years of age, inclusive.
* Body mass index (BMI) between 18 and 33 kg/m², inclusive, at screening.
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial.
* Willing to maintain current dietary supplement and non exclusionary medication use throughout the trial.
* Willing to avoid the consumption of alcohol, unusual food intake, unusual physical activity and consumption of any flatulence promoting foods 24h prior to each study visit. Failure to follow will result in rescheduled visit.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected. health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria.
* Known history of gastrointestinal disease (e.g., diverticulitis, Crohns disease, coeliac disease etc.), bariatric surgery, AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, or biliary diseases, or any condition which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or any medication which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow INQUIS health and safety policies.
* Known intolerance, sensitivity or allergy to test foods.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
* History of cancer in the prior two years, except for non-melanoma skin cancer.
* Exposure to any non-registered drug product within 30 d prior to screening.
* Self reported pregnancy or breastfeeding.
* Any history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, binge eating) diagnosed by a health professional.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | Acute response over 2 hours
  Compare the postprandial glucose incremental area under the curve response of ALLSWEET® with sucrose when taken alone or when added to sucrose.

SECONDARY OUTCOMES:
Postprandial glycemic response | Acute response over 2 hours
  Compare the postprandial glucose levels at each time point after each test meal.
Postprandial insulinemic response | Acute response over 2 hours
  Compare the postprandial insulin levels at each time point and incremental area under teh curve after each meal.

CONTACTS AND LOCATIONS:
Locations (1):
- INQUIS Clinical Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No